CLINICAL TRIAL: NCT00785785
Title: A Randomized, Open Label, Multi-center Phase III Study to Evaluate the Efficacy and Safety of Nilotinib Versus Imatinib in Adult Patients With Unresectable or Metastatic Gastrointestinal Stromal Tumors (GIST)
Brief Title: A Study of Nilotinib Versus Imatinib in GIST Patients
Acronym: ENESTg1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107G2301; 2008-004758-34 (EudraCT Number)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: Unresectable GIST; metastatic GIST; nilotinib; AMN107; imatinib; STI571
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib; Imatinib Mesylate

ARMS (2):
- Nilotinib (Experimental): nilotinib 400 mg twice a day
  Interventions: Drug: Nilotinib (AMN107)
- Imatinib (Active Comparator): imatinib 400 mg once daily
  Interventions: Drug: imatinib (STI571)

INTERVENTIONS:
Drug: Nilotinib (AMN107)
  Arms: Nilotinib
Drug: imatinib (STI571)
  Other Names: Glivec/Gleevec
  Arms: Imatinib

SUMMARY:
This study will evaluate efficacy and safety of nilotinib versus imatinib in adult patients with unresectable or metastatic gastrointestinal stromal tumors (GIST).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of GIST which is unresectable and/or metastatic and either:

   * have not received any prior anti-neoplastic therapy other than adjuvant imatinib. Note: newly diagnosed patients may have received up to 14 days of treatment with imatinib for disease management while awaiting entry to the study or
   * recurrent GIST after stopping adjuvant treatment with imatinib and no subsequent treatment with any other therapies.
2. At least one measurable site of disease on CT/MRI scan
3. Performance status ≤ 2 (capable of self-care but unable to carry out any work)
4. Normal organ, electrolyte and marrow function

Exclusion Criteria:

1. Any prior anti-neoplastic therapy with the exception of patients who have received adjuvant imatinib or patients with newly diagnosed metastatic/ unresectable GIST whose disease requires therapy while awaiting entry to the study.
2. Disease progression during adjuvant therapy with imatinib
3. History of active malignancy (other than GIST) within 10 years prior to study entry with the exception of previous or concomitant basal cell skin cancer, previous cervical carcinoma in situ.
4. Impaired cardiac function

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2009-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (155):
- United States (28):
  - Birmingham Hematology and Oncology Associates, Birmingham, Alabama
  - Northern Arizona Hematology/Oncology Associates, P.C. Dept. of No. AZ Hem-Onc, Flagstaff, Arizona
  - City of Hope National Medical Center Dept.ofCityofHopeMedicalCtr(4), Duarte, California
  - City of Hope National Medical Center Regulatory Document, Duarte, California
  - University of California San Diego - Moores Cancer Center Dept of Moores Cancer Ctr (2), La Jolla, California
  - University of California at Los Angeles GI Oncology Program, Los Angeles, California
  - Stanford University Medical Center Stanford Cancer Center, Stanford, California
  - University of Colorado Dept. of Univ. of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Centers Dept. of Rocky Mountain Cancer, Greenwood Village, Colorado
  - Washington Hospital Center Wash Hospital, Washington D.C., District of Columbia
  - Ocala Oncology Center Dept. of Ocala Oncology Center, Ocala, Florida
  - Kootenai Medical Center Dept.ofKootenai Med.Ctr., Coeur d'Alene, Idaho
  - Northwestern University Clinical Research Office (2), Chicago, Illinois
  - Dana Farber Cancer Institute Centerfor Sarcoma&BoneOncology, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center DeptofMichiganCancerCenter(6), Ann Arbor, Michigan
  - Minnesota Oncology Hematology, P.A. SC, Minneapolis, Minnesota
  - Mayo Clinic - Rochester Division of Hematology, Rochester, Minnesota
  - New York Oncology Hematology, P.C. NYOH Amsterdam, Troy, New York
  - New York Oncology Hematology, P.C. NYOH@AlbanyMedicalCenter(2), Troy, New York
  - University of Pennsylvania Medical Center CAMN107G2301, Philadelphia, Pennsylvania
  - Vanderbilt Univeristy Ingram Cancer Ctr., Nashville, Tennessee
  - Texas Oncology, P.A. Tex Onc (2), Bedford, Texas
  - Texas Oncology Wichita Falls, Dallas, Texas
  - University of Texas Southwestern Medical Center DeptofSimmons Cancer Center(3), Dallas, Texas
  - University of Texas/MD Anderson Cancer Center Dept. of MD Anderson (13), Houston, Texas
  - Cancer Care Centers of South Texas / HOAST CCC of So. TX- San Antonio(2), San Antonio, Texas
  - Tyler Cancer Center Dept.ofTylerCancerCtr. (2), Tyler, Texas
  - University of Utah / Huntsman Cancer Institute Dept.ofHuntsmanCancerInst.(3), Salt Lake City, Utah
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Austria (5):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Wels
- Brazil (4):
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (2):
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (7):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- China (5):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Pereira, Colombia
- Novartis Investigative Site, Olomouc, Czechia
- Denmark (2):
  - Novartis Investigative Site, Århus C
  - Novartis Investigative Site, Herlev
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- France (9):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (7):
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Weiden
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
- Italy (10):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Torino, TO
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
- Mexico (3):
  - Novartis Investigative Site, Chihuahua City, Chihuahua
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Mexico City, Mexico City
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Poland (2):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
- Romania (4):
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Iași
- Russia (4):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Bratislava, Slovak Republic, Slovakia
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Pretoria
- South Korea (2):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
- Spain (4):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Oviedo, Principality of Asturias
- Sweden (6):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Taiwan (4):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Linkou District
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Adana, Turkey
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Kartal
- United Kingdom (5):
  - Novartis Investigative Site, Newcastle upon Tyne, Newcastle-upon-Tyne
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
- Novartis Investigative Site, Caracas, Distrito Federal, Venezuela

REFERENCES:
- [Derived] Blay JY, Shen L, Kang YK, Rutkowski P, Qin S, Nosov D, Wan D, Trent J, Srimuninnimit V, Papai Z, Le Cesne A, Novick S, Taningco L, Mo S, Green S, Reichardt P, Demetri GD. Nilotinib versus imatinib as first-line therapy for patients with unresectable or metastatic gastrointestinal stromal tumours (ENESTg1): a randomised phase 3 trial. Lancet Oncol. 2015 May;16(5):550-60. doi: 10.1016/S1470-2045(15)70105-1. Epub 2015 Apr 14. PMID 25882987
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=717

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib First, Then Nilotinib: patients were on imatinib 400mg once daily in the core phase and then crossed over to nilotinib 400 mg twice a day in the extension phase
- Nilotinib First, Then Imatinib: patients were on nilotinib 400 mg twice a day in the core phase and then crossed over to in the extension phase imatinib 400mg once daily
Period: Core Phase up to 36 Months
Arm/Group | Imatinib First, Then Nilotinib | Nilotinib First, Then Imatinib
Started | 324 | 320
Completed | 0 | 0
Not Completed | 324 | 320
Not completed — Patients didn't receive 1st line therapy | 3 | 4
Not completed — Adverse Event | 31 | 21
Not completed — Abnormal laboratory value | 1 | 0
Not completed — Abnormal test procedure result | 2 | 2
Not completed — Withdrawal by Subject | 16 | 17
Not completed — Lost to Follow-up | 3 | 7
Not completed — Administrative problems | 3 | 3
Not completed — Death | 5 | 8
Not completed — Disease progression | 139 | 119
Not completed — Protocol deviation | 5 | 6
Not completed — Study terminated by sponsor | 116 | 133
Period: Optional Extension Phase
Arm/Group | Imatinib First, Then Nilotinib | Nilotinib First, Then Imatinib
Started | 39 (crossover extension phase was optional) | 125 (crossover extension phase was optional)
Completed | 0 | 0
Not Completed | 39 | 125
Not completed — Adverse Event | 4 | 5
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 2 | 0
Not completed — Death | 1 | 5
Not completed — Disease progression | 22 | 70
Not completed — Protocol deviation | 0 | 2
Not completed — Study terminated by sponsor | 3 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib First, Then Nilotinib | Nilotinib First, Then Imatinib | Total
Number analyzed (Participants) | 324 | 320 | 644
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.91) | 57.3 (12.63) | 57.35 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 133 | 278
  Male | 179 | 187 | 366

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to month 37
Population: Full Analysis Set (FAS) consists of all randomized patients for the Core Phase.
Measure: Median (Full Range); unit: months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 324 | 320
months | 25.9 [0 to 32.8] | 29.7 [0 to 36.1]
Statistical Analysis 1: Comparison: Nilotinib vs Imatinib; Test type: Superiority or Other; p = 0.0081, Hazard Ratio; Hazard Ratio (HR) = 1.466, 95% CI 2-sided [1.104 to 1.945]

ADVERSE EVENTS:
Groups:
- Nilotinib: Exposure to Nilotinib only
- Imatinib: Exposure to Imatinib only
- Crossover Nilotinib: exposure to imatinib and then nilotinib
- Crossover Imatinib: exposure to nilotinib and then imatinib
Arm/Group | Nilotinib | Imatinib | Crossover Nilotinib | Crossover Imatinib
Serious Adverse Events (participants affected / at risk) | 80/321 | 85/316 | 15/39 | 26/125
Other Adverse Events (participants affected / at risk) | 291/321 | 289/316 | 28/39 | 89/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=321) | Imatinib (N=316) | Crossover Nilotinib (N=39) | Crossover Imatinib (N=125)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 15 | 12 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 0 | 2
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 5 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 2 | 1 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Jejunal perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3 | 1 | 4
Asthenia (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0 | 1
Oedema mucosal (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 1 | 0
Pain (General disorders) | 0 | 0 | 2 | 1
Performance status decreased (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 6 | 0 | 3
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 4 | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 2 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 2 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cytoreductive surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0
Gastrectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Tumour excision (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=321) | Imatinib (N=316) | Crossover Nilotinib (N=39) | Crossover Imatinib (N=125)
Anaemia (Blood and lymphatic system disorders) | 38 | 61 | 7 | 20
Leukopenia (Blood and lymphatic system disorders) | 4 | 35 | 1 | 10
Neutropenia (Blood and lymphatic system disorders) | 4 | 42 | 1 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5 | 2 | 1
Eyelid oedema (Eye disorders) | 5 | 55 | 0 | 19
Lacrimation increased (Eye disorders) | 3 | 21 | 0 | 3
Periorbital oedema (Eye disorders) | 2 | 58 | 0 | 9
Abdominal distension (Gastrointestinal disorders) | 17 | 12 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 63 | 61 | 6 | 18
Abdominal pain upper (Gastrointestinal disorders) | 38 | 15 | 1 | 5
Constipation (Gastrointestinal disorders) | 49 | 24 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 46 | 106 | 2 | 17
Nausea (Gastrointestinal disorders) | 73 | 105 | 12 | 20
Stomatitis (Gastrointestinal disorders) | 10 | 14 | 2 | 1
Vomiting (Gastrointestinal disorders) | 51 | 65 | 5 | 10
Asthenia (General disorders) | 27 | 29 | 0 | 6
Face oedema (General disorders) | 5 | 43 | 0 | 13
Fatigue (General disorders) | 66 | 65 | 7 | 12
Oedema peripheral (General disorders) | 29 | 68 | 2 | 17
Pyrexia (General disorders) | 23 | 30 | 3 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 63 | 11 | 3 | 3
Nasopharyngitis (Infections and infestations) | 25 | 19 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 17 | 0 | 1
Alanine aminotransferase increased (Investigations) | 45 | 18 | 5 | 3
Amylase increased (Investigations) | 8 | 13 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 23 | 15 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 7 | 3 | 3 | 2
Blood bilirubin increased (Investigations) | 32 | 4 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 9 | 2 | 4 | 1
Haemoglobin decreased (Investigations) | 10 | 20 | 3 | 5
Lipase increased (Investigations) | 27 | 23 | 1 | 6
Neutrophil count decreased (Investigations) | 2 | 24 | 1 | 7
Weight decreased (Investigations) | 27 | 20 | 3 | 3
White blood cell count decreased (Investigations) | 3 | 21 | 0 | 11
Decreased appetite (Metabolism and nutrition disorders) | 40 | 50 | 5 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 7 | 2 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 5 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 19 | 0 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 20 | 53 | 3 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 15 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 18 | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 47 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 17 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 16 | 2 | 3
Dizziness (Nervous system disorders) | 22 | 19 | 2 | 4
Dysgeusia (Nervous system disorders) | 10 | 9 | 2 | 3
Headache (Nervous system disorders) | 54 | 24 | 5 | 2
Insomnia (Psychiatric disorders) | 21 | 20 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 21 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 21 | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 33 | 13 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 19 | 21 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 39 | 25 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 89 | 46 | 4 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.